CLINICAL TRIAL: NCT02799784
Title: A Randomized, Open-Label, 8-Week Cross-Over Study to Compare Umeclidinium/Vilanterol With Tiotropium/Olodaterol Once-Daily in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: An Efficacy Study of Umeclidinium/Vilanterol With Tiotropium/Olodaterol in COPD Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 204990
Record Dates: First submitted 2016-06-02; First posted 2016-06-15 (Estimated); Results first posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: tiotropium; COPD; olodaterol; Umeclidinium bromide; efficacy; vilanterol
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Albuterol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sequence 1: UMEC/VI 62.5/ 25 mcg (Experimental): Subjects will receive UMEC/VI 62.5/25 mcg (as one inhalation) administered QD via the ELLIPTA Inhaler for 8 weeks followed by a washout period of 3 weeks
  Interventions: Drug: UMEC/VI; Drug: Albuterol/salbutamol
- Sequence 2: TIO/OLO 5/5 mcg (Experimental): Subjects will receive TIO/OLO 5/5 mcg (as 2 inhalations of 2.5/2.5 mcg per inhalation) administered QD via the RESPIMAT inhaler for 8 weeks followed by a washout period of 3 weeks
  Interventions: Drug: TIO/OLO; Drug: Albuterol/salbutamol

INTERVENTIONS:
Drug: UMEC/VI — ELLIPTA dry powder inhaler (DPI) will contain a total of 30 doses. Each DPI will be comprised of two double-foil, laminate blister strips. Each blister of one strip will consist of 62.5 mcg of UMEC blended with lactose and magnesium stearate while each blister of other strip will consist of 25 mcg of VI blended with lactose and magnesium stearate. Each actuation of the DPI will deliver the contents of one blister from each strip simultaneously
  Arms: Sequence 1: UMEC/VI 62.5/ 25 mcg
Drug: TIO/OLO — TIO/OLO inhalation spray will be supplied as an inhalation spray delivered using a RESPIMAT inhaler. Each actuation from the RESPIMAT inhaler delivers 3.124 mcg tiotropium bromide monohydrate (equivalent to 2.5 mcg tiotropium) and 2.736 mcg olodaterol hydrochloride (equivalent to 2.5 mcg olodaterol)
  Arms: Sequence 2: TIO/OLO 5/5 mcg
Drug: Albuterol/salbutamol — Albuterol/salbutamol will be supplied as an inhalation spray via metered dose inhaler and will be issued for reversibility testing at Visit 1. Albuterol/salbutamol will be permitted throughout the study for use as-needed

SUMMARY:
The primary objective of this study is to assess the effect of umeclidinium/vilanterol (UMEC/VI) versus tiotropium/olodaterol (TIO/OLO) in subjects with moderated COPD.

This is a multicentre, randomized, open label, 2 period crossover complete block design study.

Eligible subjects, who complete a 2-week run-in period, will be randomized to receive a sequence consisting of UMEC/VI inhalation powder (62.5/25 microgram [mcg] once-daily [QD]) administered as 1 inhalation via the ELLIPTA® Inhaler and TIO/OLO 5/5 mcg inhalation spray administered as 2 inhalations via the RESPIMAT® inhaler, for 8 weeks each. This will be followed by a 3-week washout period and one-week follow-up period. The total duration of subject participation in the study will be approximately 22 weeks.

ELLIPTA is a registered trademark of the GlaxoSmithKline group of companies. RESPIMAT is a registered trademark of Boehringer Ingelheim.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients of either sex, 40 years of age or older at Visit 1, and with a diagnosis of chronic obstructive pulmonary disease (COPD) defined by the American Thoracic Society/European Respiratory Society (ERS)
* A signed and dated written informed consent prior to study participation
* A female is eligible to enter and participate in the study if she is not pregnant (as confirmed by a negative urine human chorionic gonadotrophin [hCG] test); not lactating; and of non-reproductive potential (i.e., physiologically incapable of becoming pregnant, including any female who is post-menopausal or surgically sterile), which is defined as pre-menopausal females with one of the following: documented tubal ligation; documented hysteroscopic tubal occlusion procedure with follow-up confirmation of bilateral or tubal occlusion ; hysterectomy; documented bilateral oophorectomy.

Postmenopausal is defined as 12 months of spontaneous amenorrhea in questionable cases a blood sample with simultaneous follicle stimulating hormone (FSH) and estradiol levels consistent with menopause (refer to laboratory reference ranges for confirmatory levels). Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of post-menopausal status prior to study enrolment OR

* A female of reproductive potential, has a negative pregnancy test at screening, and agrees to one of the methods below in the GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in Females of Reproductive Potential (FRP) requirements from methods used consistently and correctly (i.e., in accordance with the local approved product label and per study investigator discretion and the instructions of the physician from 30 days prior to the first dose of study medication and until to follow-up contact):

GSK Modified List of Highly Effective Methods for Avoiding Pregnancy in FRP (this list does not apply to FRP with same sex partners, when this is their preferred and usual lifestyle or for subjects who are and will continue to be abstinent from penile-vaginal intercourse on a long term and persistent basis).

* Contraceptive subdermal implant that meets the standard operating procedure (SOP) effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Intrauterine device or intrauterine system that meets the SOP effectiveness criteria including a <1% rate of failure per year, as stated in the product label
* Oral Contraceptive, either combined or progestogen alone
* Injectable progestogen
* Contraceptive vaginal ring
* Percutaneous contraceptive patches
* Male partner sterilization with documentation of azoospermia prior to the female subject's entry into the study, and this male is the sole partner for that subject.

These allowed methods of contraception are only effective when used consistently, correctly and in accordance with the product label. The investigator is responsible for ensuring that subjects understand how to properly use these methods of contraception

* Current or former cigarette smokers with a history of cigarette smoking of >=10 pack-years. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 1. Pipe and/or cigar use cannot be used to calculate pack-year history.
* A pre and post-albuterol/salbutamol forced expiratory volume in one second (FEV1)/Forced Vital Capacity ratio of <0.70 and a post-albuterol/salbutamol FEV1 of <=70% to >=50 % of predicted normal values at Visit 1. Predicted values will be based upon the ERS' Global Lung Function Initiative
* A score of >=2 on the Modified Medical Research Council Dyspnea Scale at Visit 1

Exclusion Criteria:

* Women who are pregnant or lactating or are planning on becoming pregnant during the study
* A current diagnosis of asthma
* Subjects with alpha-1 antitrypsin deficiency as the underlying cause of COPD
* Subjects with active tuberculosis are excluded. Subjects with other respiratory disorders (e.g. clinically significant: bronchiectasis, sarcoidosis, lung fibrosis, pulmonary hypertension, interstitial lung diseases) are excluded if these conditions are the primary cause of their respiratory symptoms.
* Any subject who is considered unlikely to survive the duration of the study period or has any rapidly progressing disease or immediate life-threatening illness (e.g. cancer). In addition, any subject who has any other condition (e.g. neurological condition) that is likely to affect respiratory function should not be included in the study
* Current active liver or biliary disease (with the exception of Gilbert's syndrome or asymptomatic gallstones or otherwise stable chronic liver disease per investigator assessment
* Investigational Product should be used with caution in subjects with severe cardiovascular disease. In the opinion of the investigator, use should only be considered if the benefit is likely to outweigh the risk in conditions such as:

Myocardial infarction or unstable angina in the last 6 months Unstable or life threatening cardiac arrhythmia requiring intervention in the last 3 months New York Heart Association Class IV heart failure

* Any history of allergy or hypersensitivity to any anticholinergic/muscarinic receptor antagonist, sympathomimetic, lactose/milk protein or magnesium stearate
* Subjects with medical conditions such as narrow-angle glaucoma, urinary retention, prostatic hypertrophy, or bladder neck obstruction should be excluded unless, in the opinion of the study physician, the benefit outweighs the risk
* Hospitalization for COPD or pneumonia within 12 weeks prior to Visit 1. Pneumonia and/or moderate or severe COPD exacerbation that has not resolved at least 14 days prior to Screening (V1) and at least 30 days following the last dose of oral/systemic corticosteroids (if applicable).
* Other respiratory tract infections that have not resolved at least 7 days prior to Screening (V1).
* Subjects with lung volume reduction surgery (including procedures such as endobronchial valves) within the 12 months prior to Screening (V1).
* The Investigator will determine the clinical significance of each abnormal electrocardiogram finding in relation to the subject's medical history and exclude subjects who would be at undue risk by participating in the trial
* Unable to withhold albuterol/salbutamol for the 4-hour (h) period required prior to spirometry testing at each study visit
* Use of the pre-defined medications according to the pre-defined defined time intervals prior to Screening (Visit 1)
* Use of long-term oxygen therapy described as resting oxygen therapy >3 liter (L)/minute (min) at screening. (Oxygen use <=3 L/min flow is not exclusionary, and patients may adjust oxygen levels as needed during the study.)
* Regular use (prescribed for daily/ regular use, not for as-needed use) of short-acting bronchodilators (e.g. albuterol/salbutamol).
* Participation in the acute phase of a pulmonary rehabilitation program within 4 weeks prior to Screening (Visit 1). Subjects who are in the maintenance phase of a pulmonary rehabilitation program are not excluded
* A known or suspected history of alcohol or drug abuse within 2 years prior to Screening (Visit 1) that in the opinion of the investigator would prevent the subject from completing the study procedures
* Is an investigator, sub-investigator, study coordinator, employee of a participating investigator or study site, or immediate family member of the aforementioned that is involved in this study
* In the opinion of the investigator, any subject who is unable to read and/or would not be able to complete a questionnaire.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Actual)
Dates: Start 2016-07-14 (Actual); Primary Completion 2017-04-27 (Actual); Study Completion 2017-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- United States (9):
  - GSK Investigational Site, Clearwater, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, St Louis, Missouri
  - GSK Investigational Site, Medford, Oregon
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Greenville, South Carolina
  - GSK Investigational Site, Spartanburg, South Carolina
  - GSK Investigational Site, Richmond, Virginia
  - GSK Investigational Site, Morgantown, West Virginia
- Germany (7):
  - GSK Investigational Site, Frankfurt am Main, Hesse
  - GSK Investigational Site, Neu-Isenburg, Hesse
  - GSK Investigational Site, Hanover, Lower Saxony
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Jerichow, Saxony-Anhalt
  - GSK Investigational Site, Magdeburg
- Spain (7):
  - GSK Investigational Site, Marbella - Málaga, Andalusia
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Girona
  - GSK Investigational Site, Loja/ Granada
  - GSK Investigational Site, Mérida (Badajoz)
  - GSK Investigational Site, Ponferrada (León)
  - GSK Investigational Site, Valladolid
- United Kingdom (11):
  - GSK Investigational Site, Cheadle, Cheshire
  - GSK Investigational Site, Chesterfield, Derbyshire
  - GSK Investigational Site, Romford, Essex
  - GSK Investigational Site, Manchester, Greater Manchester
  - GSK Investigational Site, Salford, Greater Manchester
  - GSK Investigational Site, Northwood, Middlesex
  - GSK Investigational Site, Addlestone, Surrey
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Chippenham
  - GSK Investigational Site, Sidcup, Kent
  - GSK Investigational Site, Swinton

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Alcazar Navarrete B, Boucot I, Naya I, Tombs L, Lipson DA, Compton C, Sousa AR, Feldman G. Umeclidinium/Vilanterol Versus Tiotropium/Olodaterol in Maintenance-Naive Patients with Moderate Symptomatic Chronic Obstructive Pulmonary Disease: A Post Hoc Analysis. Pulm Ther. 2018 Dec;4(2):171-183. doi: 10.1007/s41030-018-0057-7. Epub 2018 Jun 20. PMID 32026389
- [Derived] Feldman GJ, Sousa AR, Lipson DA, Tombs L, Barnes N, Riley JH, Patel S, Naya I, Compton C, Alcazar Navarrete B. Comparative Efficacy of Once-Daily Umeclidinium/Vilanterol and Tiotropium/Olodaterol Therapy in Symptomatic Chronic Obstructive Pulmonary Disease: A Randomized Study. Adv Ther. 2017 Nov;34(11):2518-2533. doi: 10.1007/s12325-017-0626-4. Epub 2017 Nov 1. PMID 29094315
- See also: IPD for this study will be made available via the Clinical Study Data Request site. — https://clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This is a multicenter, randomized, open label, 2 period crossover complete block design study. Participants (par.) with Chronic Obstructive Pulmonary Disease (COPD) were enrolled across 4 countries: Germany, Spain, the United Kingdom and the United States.
Pre-assignment Details: Study consisted of a run-in period of approximately 2 weeks followed by two 8-week treatment periods with a washout of approximately 3 weeks. The total duration of the study was approximately 22 weeks including follow-up. A total of 443 par. were screened, of which 236 par. were randomized (207 par. were pre-screen, screen and run-in failures).
Groups:
- UMEC/VI Followed by TIO/OLO: In this 2-way crossover study, eligible participants were administered Umeclidinium/Vilanterol (UMEC/VI) 62.5/25 microgram (mcg) (as one inhalation) once-daily (QD) via ELLIPTA Inhaler for 8 weeks in TP1. It was followed by a washout period of 3 weeks. Par. received Tiotropium/Olodaterol (TIO/OLO) 5/5 mcg inhalation spray as 2 inhalations of 2.5/2.5 mcg each via the RESPIMAT® inhaler for 8 weeks in TP2. Albuterol/salbutamol was supplied as an inhalation spray via metered dose inhaler throughout the study for use as-needed
- TIO/OLO Followed by UMEC/VI: In this 2-way crossover study, eligible participants were administered TIO/OLO 5/5 mcg inhalation spray as 2 inhalations of 2.5/2.5 mcg each via the RESPIMAT® inhaler for 8 weeks in TP1. It was followed by a washout period of 3 weeks. Par. received UMEC/VI 62.5/25 mcg (as one inhalation) QD via ELLIPTA Inhaler for 8 weeks in TP2. Albuterol/salbutamol was supplied as an inhalation spray via metered dose inhaler throughout the study for use as-needed
Period: Treatment Period 1 (TP1- 8 Weeks)
Arm/Group | UMEC/VI Followed by TIO/OLO | TIO/OLO Followed by UMEC/VI
Started | 117 | 119
Completed | 111 | 118
Not Completed | 6 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 0
Period: Washout Period (3 Weeks)
Arm/Group | UMEC/VI Followed by TIO/OLO | TIO/OLO Followed by UMEC/VI
Started | 111 | 118
Completed | 111 | 118
Not Completed | 0 | 0
Period: Treatment Period 2 (TP2 - 8 Weeks)
Arm/Group | UMEC/VI Followed by TIO/OLO | TIO/OLO Followed by UMEC/VI
Started | 111 | 118
Completed | 110 | 115
Not Completed | 1 | 3
Not completed — Adverse Event | 0 | 1
Not completed — Par. reached protocol stopping criteria | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- All Treatment Combined: In this 2-way crossover study, eligible participants were randomized to receive UMEC/VI inhalation powder 62.5/25 mcg QD administered as 1 inhalation via the ELLIPTA® Inhaler and TIO/OLO 5/5 mcg inhalation spray administered as 2 inhalations via the RESPIMAT® inhaler in 8-week TP1 and TP2 per randomization. This was separated by a 3-week washout period. Albuterol/salbutamol was supplied as an inhalation spray via metered dose inhaler throughout the study for use as-needed
Arm/Group | All Treatment Combined
Number analyzed (Participants) | 236
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 142
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African Heritage | 13
  White - White/Caucasian/European Heritage | 223

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second (FEV1) at Week 8
Description: FEV1 is a measure of lung function and is defined as the maximal amount of air that can be forcefully exhaled in one second. Trough FEV1 was defined as 23 and 24 hour post-dose FEV1 measurements. All par. in the Intent To Treat (ITT) Population who were not identified as full protocol deviators were included in Per-Protocol (PP) Population. ITT Population, comprised of all randomized subjects, who received at least one dose of study medication.
Time Frame: Week 8
Population: Per Protocol Population
Measure: Least Squares Mean (Standard Error); unit: Liters
Groups:
- Umeclidinium/Vilanterol 62.5/25 mcg: Eligible par. were administered Umeclidinium/Vilanterol (UMEC/VI) 62.5/25 mcg (as one inhalation) once-daily (QD) via the ELLIPTA Inhaler for 8 weeks followed by a washout period of 3 weeks in period-1 or 2 as per randomization. Albuterol/salbutamol was supplied as an inhalation spray via metered dose inhaler throughout the study for use as-needed
- Tiotropium/Olodaterol 5/5 mcg: Eligible par. were administered Tiotropium/Olodaterol (TIO/OLO) 5/5 mcg inhalation spray as 2 inhalations of 2.5/2.5 mcg each via the RESPIMAT® inhaler for 8 weeks followed by a washout period of 3 weeks in period-1 or 2 as per randomization. Albuterol/salbutamol was supplied as an inhalation spray via metered dose inhaler throughout the study for use as-needed
Arm/Group | Umeclidinium/Vilanterol 62.5/25 mcg | Tiotropium/Olodaterol 5/5 mcg
Number analyzed (Participants) | 202 | 192
Liters | 1.745 (0.0131) | 1.692 (0.0135)
Statistical Analysis 1: Comparison: Umeclidinium/Vilanterol 62.5/25 mcg vs Tiotropium/Olodaterol 5/5 mcg; Test type: Non-Inferiority — If the lower bound of the two-sided 95% confidence interval around the (UMEC/VI 62.5/25 mcg versus TIO/OLO 5/5 mcg) treatment difference is above -50 milliliter then UMEC/VI 62.5/25 mcg was to be considered non-inferior to TIO/OLO 5/5 mcg; p < 0.001, Mixed Models Analysis; Mean Difference (Final Values) = 0.053, 95% CI 2-sided [0.026 to 0.080]

ADVERSE EVENTS:
Time Frame: On-therapy Serious Adverse Events (SAEs) and non-SAEs were collected from the start of study treatment and until follow up visit (Week 22).
Description: On-therapy SAEs and non-SAEs are reported for ITT Population, comprised of all randomized participants, who received at least one dose of study medication
Arm/Group | Umeclidinium/Vilanterol 62.5/25 mcg | Tiotropium/Olodaterol 5/5 mcg
All-Cause Mortality (participants affected / at risk) | 0/235 | 0/230
Serious Adverse Events (participants affected / at risk) | 3/235 | 2/230
Other Adverse Events (participants affected / at risk) | 19/235 | 21/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 mcg (N=235) | Tiotropium/Olodaterol 5/5 mcg (N=230)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Catheter site haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umeclidinium/Vilanterol 62.5/25 mcg (N=235) | Tiotropium/Olodaterol 5/5 mcg (N=230)
Viral upper respiratory tract infection (Infections and infestations) | 11 (11) | 14 (15)
Upper respiratory tract infection (Infections and infestations) | 8 (8) | 7 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2016-03-29): https://cdn.clinicaltrials.gov/large-docs/84/NCT02799784/Prot_000.pdf
  • Statistical Analysis Plan (2017-05-26): https://cdn.clinicaltrials.gov/large-docs/84/NCT02799784/SAP_001.pdf